CLINICAL TRIAL: NCT02024555
Title: Investigation of the Efficacy of Antimycobacterial Therapy on Pulmonary Sarcoidosis Phase II Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Phase II Investigation of Antimycobacterial Therapy on Progressive, Pulmonary Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Wonder Drake, Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HL117074 (NIH); R01HL117074-01 (NIH)
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Sarcoidosis; Antimycobacterial Therapy
MeSH Terms: conditions — Sarcoidosis | interventions — Levofloxacin; Ethambutol; Azithromycin; Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin (Active Comparator): Levofloxacin 500mg po QD; Ethambutol 1200mg po QD; Azithromycin 250 mg po QD; Rifampin 600mg po QD or Rifabutin 300mg po QD
  Interventions: Drug: Levofloxacin; Drug: Ethambutol; Drug: Azithromycin; Drug: Rifampin
- Placebo (Placebo Comparator): Riboflavin will be used for rifampin; encapsulated microcrystalline cellulose will be used to replace the levofloxacin, ethambutol and azithromycin.
  The pill count will be the same as the comparator regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levofloxacin
  Other Names: Levaquin
  Arms: Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin
Drug: Ethambutol
  Arms: Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin
Drug: Azithromycin
  Other Names: Z-pack
  Arms: Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin
Drug: Rifampin
  Other Names: Rifadin, Rimactane
  Arms: Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin
Drug: Placebo — This will serve as a placebo to the antibiotics used in antimycobacterial therapy.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to investigate the efficacy and safety of oral antimycobacterial therapy in patients with confirmed progressive pulmonary sarcoidosis. We suspect that the CLEAR regimen will improve the absolute FVC percent predicted in chronic pulmonary sarcoidosis participants.

DETAILED DESCRIPTION:
Primary Objective: To assess the efficacy and safety of oral CLEAR therapy in patients with confirmed progressive pulmonary sarcoidosis.

Hypothesis: The CLEAR regimen will improve the absolute FVC percent predicted in chronic pulmonary sarcoidosis participants by augmenting T cell responses through the normalization of p56Lck expression and IL-2 production.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoidosis as defined by the ATS/ERS/WASOG statement on sarcoidosis as defined by the clinical presentation consistent with sarcoidosis, as well as biopsy demonstrating granulomas, and no alternative for the cause of the granulomas, such as tuberculosis for at least one year prior to randomization.
2. Evidence of disease progression as defined by at least one of the following three criteria:

   Decline of absolute percent predicted of FVC (FVC ≥45% or higher of predicted value) or DLCO of at least 5% on serial measurements (DLCO range >35%, if measured); Radiographic progression in chest imaging on side by side comparison; Change in dyspnea score, as measured by Transition Dyspnea Index (TDI); Positive peripheral immune responses to ESAT-6 as a biomarker of response to CLEAR regimen.
3. Possess evidence of parenchymal or nodal disease on chest radiograph.

Exclusion Criteria:

1. Inability to obtain consent
2. Age less than 18 years
3. Female participants of childbearing potential not willing to use one of the following methods of birth control for the duration of the study and 90 days after study completion: condoms, sponge, foams, jellies, diaphragm, non-hormonal intrauterine device, a vasectomized sole partner or abstinence. Note: Oral contraceptive pills are not effective birth control when taking rifamycin. A negative urine pregnancy test at screening visit if female of childbearing potential
4. FVC predicted value is < 45%.
5. End-stage fibrotic pulmonary disease.
6. Significant underlying liver disease.
7. Allergy or intolerance to any of the antibiotics within the CLEAR regimen.
8. Allergy or intolerance to albuterol
9. Poor venous access for obtaining blood samples
10. History of active tuberculosis, close contact with a person with active tuberculosis within the 6 months prior to the screening visit or has a positive PPD.
11. Significant disorder, other than sarcoidosis, that would complicate the treatment evaluation, (such as respiratory, cardiac, neurologic, musculoskeletal or seizure disorders)
12. Use of an investigational drug within 30 days prior to screening or within 5 half-lives of the agent, whichever is longer.
13. Currently receiving >40mg prednisone.
14. ALT or AST >5 times upper limit of normal (ULN)
15. Leukopenia, as defined by WBC <3.0 cells/mm3 or absolute neutrophil count <1000
16. Breast feeding.
17. Color perception impairment as defined by the inability to differentiate colors per personal history or history of optic neuritis from any cause, including from sarcoidosis.
18. If patient is on immunomodulators, they must be on regimen for ≥ 3-month period and on a stable dose for > 4 weeks.
19. Family or personal history of long QT interval
20. Most recent nuclear medicine scan or echocardiogram (if done), demonstrating cardiac ejection fraction <35%
21. Participant has persistent or active infection(s) requiring hospitalization or treatment with antibiotics, antiretrovirals, or antifungals within 30 days prior to baseline. Minocycline and doxycycline are not considered antibiotics when used to treat sarcoidosis.
22. Any significant finding in the patient's medical history or physical or psychiatric exam prior to or after randomization that, in the opinion of the investigator, would affect patient safety or compliance or ability to deliver the study drug according to protocol.
23. On medications that interact with the antibiotics of the CLEAR regimen
24. History of or receiving treatment for pulmonary hypertension. Receiving biologic medication within the 6 months prior to screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-03; Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wonder Drake, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (6):
- United States (6):
  - Albany Medical Center, Albany, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University School of Medicine, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 446 participants were screened but only 97 participants met inclusion/exclusion and were randomized.
Groups:
- Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin: Levofloxacin 500mg po QD; Ethambutol 1200mg po QD; Azithromycin 250 mg po QD; Rifampin 600mg po QD or Rifabutin 300mg po QD
  Levofloxacin
  Ethambutol
  Azithromycin
  Rifampin
- Placebo: Riboflavin will be used for rifampin; encapsulated microcrystalline cellulose will be used to replace the levofloxacin, ethambutol and azithromycin.
  The pill count will be the same as the comparator regimen.
  Placebo: This will serve as a placebo to the antibiotics used in antimycobacterial therapy.
Period: Overall Study
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Started | 49 | 48
Completed (includes those who did not complete the entire study drug regime but did complete study visits) | 43 | 46
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (9.8) | 54.5 (10.4) | 54.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 47
  Male | 29 | 21 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 48 | 46 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 15 | 13 | 28
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
Weight [Mean (Standard Deviation); unit: kilograms] | 92.78 (24.45) | 97.54 (21.99) | 95.19 (23.24)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 79.59 (17.7) | 76.19 (11.66) | 77.91 (13.33)
6 minute walk test [Mean (Standard Deviation); unit: meters] — The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes
  meters | 416.25 (140.69) | 416.49 (105.16) | 416.33 (123.55)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Predicted Absolute Forced Vital Capacity (FVC) in Participants With Pulmonary Sarcoidosis, Comparing Baseline With Performance After Completion of 16 Weeks of Therapy.
Description: Change in percent predicted absolute forced vital capacity (FVC) in participants with pulmonary sarcoidosis, comparing baseline with performance after completion of 16 weeks of therapy. This will involve comparing sarcoidosis and placebo after 16 weeks of therapy.
Time Frame: Baseline to 16 weeks
Population: Only 43 participants in each arm completed this measure
Measure: Mean (Standard Deviation); unit: percentage predicted absolute FVC
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 43 | 43
percentage predicted absolute FVC | 0.35 (6.76) | 0.17 (7.2)

2. Secondary Outcome: Radiographic Improvement in Sarcoidosis Lung Disease by Frontal Chest X-ray .
Description: Radiographic improvement in sarcoidosis lung disease by frontal chest x-ray . Local investigators will score chest x-rays.
Time Frame: Baseline and 16 weeks
Population: The outcome was not completed due to lack of funds for radiology services.
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Six Minute Walk, Distance in Meters
Description: The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.
Time Frame: Baseline, 4, 8, and 16 and 24 weeks
Population: Week 24 assessment was optional. Not all participants completed the 6 minute walk test.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 48 | 48
meters
  Baseline | 416.25 (140.69) | 416.41 (105.15)
  Week 4: number analyzed (Participants) | 23 | 27
  Week 4 | 432.65 (155.5) | 428.35 (92.36)
  Week 8: number analyzed (Participants) | 24 | 23
  Week 8 | 451.59 (146.12) | 420.21 (93.9)
  Week 16: number analyzed (Participants) | 39 | 41
  Week 16 | 440.37 (137.08) | 430.85 (111.96)
  Week 24: number analyzed (Participants) | 19 | 16
  Week 24 | 444.68 (165.09) | 425.18 (104.95)

4. Secondary Outcome: Change in Oxygen Saturation
Description: measured using pulse oximetry
Time Frame: Baseline, 4, 8, and 16 and 24 weeks
Population: not all participants completed the measure and it was not recorded at week 24
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 49 | 48
percentage of oxygen saturation
  Baseline to week 4: number analyzed (Participants) | 23 | 27
  Baseline to week 4 | 0.39 (3.33) | -0.85 (1.95)
  Baseline to week 8: number analyzed (Participants) | 25 | 23
  Baseline to week 8 | -0.12 (2.95) | -0.43 (3.31)
  Baseline to week 16: number analyzed (Participants) | 43 | 43
  Baseline to week 16 | 2.54 (14.80) | -0.46 (3.79)
  Baseline to week 24: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Level of Dyspnea
Description: Outcome measure if a composite
Time Frame: Baseline, 4, 8 and 16 weeks
Population: this measure was not administered
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in the Saint George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction.
  Scores range from 0 to 100, with higher scores indicating more limitations.
  A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing.
Time Frame: Baseline and 16 weeks
Population: questionnaire was only administered at baseline and 16 weeks and not all participants completed the questionnaire at week 16
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 41 | 39
score on a scale | -2.23 (11.9) | -6.30 (9)

7. Secondary Outcome: Fatigue Assessment Scale (FAS).
Description: The FAS is a 10-item general fatigue questionnaire to assess fatigue. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
Time Frame: Baseline, 4, 8, 16 and 24 weeks
Population: The FAS was not administered to participants.
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in the King's Sarcoidosis Questionnaire (KSQ) for the Assessment of Health Status;
Description: The KSQ is a free, online questionnaire to be filled out by sarcoidosis patients. The questionnaire takes around 10 minutes and is split into 5 sections; general health status, lungs, medication, skin and eyes. There are 29 questions in total, however some questions may not be answered (depending on the type of sarcoidosis affected). Each question asks patients to rate how they feel about many different aspects of their life, for instance how much pain they are in or how difficult they find everyday tasks. Information provided is confidential. Results are given as a number between 1-100 with higher numbers indicating better health.
Time Frame: Baseline and 16 weeks
Population: KSQ was not administered to participants.
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Adverse Events
Description: Safety profile of regimen as evidenced by the number of adverse events
Time Frame: 24 weeks
Measure: Number; unit: number of events
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 49 | 48
number of events
  Serious Adverse Events | 4 | 3
  Non-Serious Adverse Events | 24 | 16

10. Secondary Outcome: FEV1%
Description: FEV1% was measure pre and post 6 minute walk test
Time Frame: Baseline, 4, 8, and 16 and 24 weeks
Population: Week 24 assessment was optional. Not all participants completed all measurements
Measure: Mean (Standard Error); unit: Percentage of predicted FEV1
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 49 | 48
Percentage of predicted FEV1
  Baseline pre | 69.11 (17.23) | 67.45 (17.85)
  Baseline post: number analyzed (Participants) | 45 | 47
  Baseline post | 69.97 (17.01) | 73.81 (18.91)
  4 weeks pre: number analyzed (Participants) | 23 | 26
  4 weeks pre | 71.57 (17.31) | 69.56 (20.52)
  4 weeks post: number analyzed (Participants) | 21 | 25
  4 weeks post | 71.96 (16.46) | 73.81 (18.91)
  8 weeks pre: number analyzed (Participants) | 25 | 23
  8 weeks pre | 69.30 (17.22) | 73.71 (19.01)
  8 weeks post: number analyzed (Participants) | 22 | 22
  8 weeks post | 70.36 (17.62) | 74.3 (19.05)
  16 weeks pre: number analyzed (Participants) | 43 | 43
  16 weeks pre | 69.88 (16.5) | 68.27 (20.17)
  16 weeks post: number analyzed (Participants) | 40 | 41
  16 weeks post | 71.39 (18.33) | 70.41 (20.03)
  24 weeks pre: number analyzed (Participants) | 19 | 17
  24 weeks pre | 72.22 (17.73) | 63.27 (20.17)
  24 weeks post: number analyzed (Participants) | 19 | 17
  24 weeks post | 73.09 (18.333) | 66.27 (19.78)

11. Secondary Outcome: Failure of Standard Therapy
Description: We will assess how many subjects in either arm need escalation of their standard regimen (ie increase in prednisone) during the 16 weeks.
Time Frame: Baseline to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 43 | 48
Participants | 3 | 2

12. Secondary Outcome: Abnormal Lab Values
Description: Safety profile of regimen as evidenced by the number of abnormal lab values classified as Adverse Events
Time Frame: baseline to 16 weeks
Measure: Number; unit: participants
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
Number analyzed (Participants) | 49 | 48
participants
  low platelet count | 1 | 0
  low WBC count | 5 | 0
  elevated glucose | 3 | 2
  low glucose | 1 | 1

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/49 | 3/48
Other Adverse Events (participants affected / at risk) | 24/49 | 16/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin (N=49) | Placebo (N=48)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Neurosarcoidosis (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis from Abcess (Infections and infestations) | 0 (0) | 1 (1)
post-operative infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant Levaquin, Ethambutol, Azithromycin and Rifampin (N=49) | Placebo (N=48)
Low Platelet count (Blood and lymphatic system disorders) | 1 | 0
Low WBC Count (Blood and lymphatic system disorders) | 1 | 0
leukopenia (Blood and lymphatic system disorders) | 1 | 0
WBC Low (Blood and lymphatic system disorders) | 1 | 0
Low WBC (Blood and lymphatic system disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
Loss of Hearing in Right Ear (Ear and labyrinth disorders) | 0 | 1
Elevated Glucose (Endocrine disorders) | 1 | 0
hypoglycemia (Endocrine disorders) | 1 | 0
Worsening Glucose (Endocrine disorders) | 0 | 1
hypoglycemia (Endocrine disorders) | 0 | 1
elevated glucose (Endocrine disorders) | 0 | 1
Floater/Blurry Vision (Eye disorders) | 1 | 0
Eyes red & draining (Eye disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 1 | 0
loss of appetite (Gastrointestinal disorders) | 1 | 0
weakness (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
diarrhea/loose stool (Gastrointestinal disorders) | 1 | 0
Nausea, Vomiting, Diarrhea (Gastrointestinal disorders) | 1 | 0
Nauseated, Vomiting & Diarrhea (Gastrointestinal disorders) | 1 | 0
nausea, vomitting, diarrhea (Gastrointestinal disorders) | 1 | 0
Surgey (Appendectomy) (Gastrointestinal disorders) | 0 | 1
Nausea & Diarrhea (Gastrointestinal disorders) | 0 | 1
Diarrhea, loss of appetite, (Gastrointestinal disorders) | 0 | 1
Fever, Nausea, Chills (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
increase in hair loss (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Insomnia (General disorders) | 1 | 0
Urine Color change (General disorders) | 1 | 0
Tiredness/Fatigue (General disorders) | 1 | 0
flu-like symptoms (chills, aches, fatigue) (General disorders) | 1 | 0
Dehydration (General disorders) | 1 | 0
Hospitalization (General disorders) | 1 | 0
Right Upper Quadant Pain (General disorders) | 1 | 0
fever, chills (General disorders) | 1 | 0
Pruritus (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Tiredness (General disorders) | 0 | 1
Hard to swallow (General disorders) | 0 | 1
elevated LFTs (Hepatobiliary disorders) | 1 | 0
yeast infection (Infections and infestations) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Yeast Infection, (Urine Urgency, Fever, Joint Aches) (Infections and infestations) | 1 | 0
Foot Abscess (Infections and infestations) | 0 | 1
Sinus Infection (Infections and infestations) | 0 | 1
Reaction to medication (Injury, poisoning and procedural complications) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
broken foot and fibula (Injury, poisoning and procedural complications) | 0 | 1
joint pain and achiness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Stiffiness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
muscle/flank/joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
confusion (Nervous system disorders) | 1 | 0
depression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety, Insomnia (Psychiatric disorders) | 1 | 0
Kidney stone pain (Renal and urinary disorders) | 0 | 1
SOB/Fatigue (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough, fever chills, pain with breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Elevated Glucose (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus blockage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
cough, wheeze, congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT02024555/Prot_SAP_000.pdf